CLINICAL TRIAL: NCT05672225
Title: Effectiveness of Two-channel Intravenous Patient-controlled Analgesia With Dexmedetomidine on Postoperative Opioid Consumption After Major Laparoscopic Abdominal Surgery
Brief Title: Two-channel IV-PCA With Dexmedetomidine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seok Kyeong Oh, Associate Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022GR0414
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Analgesia, Patient-Controlled; Dexmedetomidine
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Continuous channel: normal saline 100ml, 2ml/h (fixed rate) Selector & Bolus channel: fentanyl 20mcg/kg (Total 50ml with normal saline), bolus 1ml/10min lock-out
  Interventions: Drug: Control
- Dexmedetomidine group (Experimental): Continuous channel: dexmedetomidine 10mcg/kg (Total 100ml with normal saline), 2ml/h (fixed rate) Selector & Bolus channel: fentanyl 20mcg/kg (Total 50ml with normal saline), bolus 1ml/10min lock-out
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.2mcg/kg/hr (2ml/hr) administration via continuous channel in the experimental group
  Arms: Dexmedetomidine group
Drug: Control — Normal saline 2ml/hr administration via continuous channel in the experimental group
  Arms: Control group

SUMMARY:
Dexmedetomidine was administered in the 'selector' channel and fentanyl in the 'basic & bolus' channel of dual channel intravenous patient-controlled analgesia (IV-PCA) and the amount of opioid consumption was compared. In addition, intensity of pain, postoperative nausea/vomiting, and postoperative delirium was evaluated.

DETAILED DESCRIPTION:
Bellomic® (Cebika, Uiwang-si, Gyeonggi-do, South Korea), a new IV-PCA device consisting of two separate drug pump channels, can be used in various ways and is expanding its scope of use. Unlike conventional IV-PCA devices, which have been used to mix and administer all drugs in one channel, the device can inject drugs separately in two channels. One channel (Selector & Bolus) allows the patient to control whether to take additional bolus medication by pressing the button with adjustable continuous infusion, while the other channel (Continuous) allows constant rate continuous infusion.

Dexmedetomidine is a selective alpha-2 agonist, which is widely used in intensive care unit management, surgery, and various procedures because it has the advantage of less respiratory suppression along with sedation/anesthesia and pain effects. It has been previously reported that postoperative pain, morphine usage, and nausea/vomiting can be reduced when used during/after surgery in addition to general anesthetic drugs. However, in terms of major abdominal surgery, there is no research related to the use of dexmedetomidine after surgery, even though a large amount of opioid agents are required due to severe acute pain.

Thus, the investigators planned a randomized controlled trial to investigate the effectiveness dexmedetomidine using dual-chamber IV-PCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was scheduled for laparoscopic major abdominal surgery (Gastrectomy, Hepatectomy, Colectomy, Pancreatectomy) under general anesthesia
* Aged ≥ 20 years old

Exclusion Criteria:

* Body mass index ≥35 kg/m2
* American Society of Anesthesiologists physical status > 3
* Severe cardiovascular disorder
* Severe liver or renal dysfunction
* Preoperative dyspnea
* Contraindication to dexmedetomidine (preoperative severe bradycardia (Heart rate <50), atrioventricular block, allergy to dexmedetomidine)
* Preoperative use of opioid, anticonvulsant, antidepressant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fentanyl consumption during 24 hours | 24 hours after surgery
  Cumulative consumption of fentanyl during 24 hours

SECONDARY OUTCOMES:
Additional analgesic consumption at post-anesthesia care unit | 1 hour after surgery
  Opioid, NSAID, or acetaminophen consumption
Fentanyl consumption during 1,6,48 hours | 1,6,24,48 hours after surgery
  Cumulative consumption of fentanyl during 1,6,48 hours
Pain scores at 1,6,24,48 hours | 1,6,24,48 hours after surgery
  11-pointed numerical rating scale pain score (0 [no pain]-10 [Extreme pain])
Rescue analgesic consumption at 1,6,24,48 hours | 1,6,24,48 hours after surgery
  Additional opioid, NSAID, or acetaminophen consumption
Adverse events during 1,6,24,48 hours | 1,6,24,48 hours after surgery
  Nausea, vomiting, hypotension, sedation, respiratory depression, pruritus
Delirium during 1,6,24,48 hours | 1,6,24,48 hours after surgery
  Confusion assessment method (CAM)-evaluated delirium
Satisfaction score at 24 hours | 24 hours after surgery
  Satisfaction score evaluated with quality of recovery (QoR)-15 (0[poor] to 10[excellent]), 7-pointed Likert scale (1 [very dissatisfied]- 7[very satisfied])

CONTACTS AND LOCATIONS:
Overall Officials: Seok Kyeong Oh, M.D., Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No